CLINICAL TRIAL: NCT06681363
Title: Creation of a Biocollection of Patients with Acute Myeloid Leukemia (AML) or Lymphoid Leukemia (ALL) or High-risk Myelodysplastic Syndrome (MDS) Monitored At the Nantes University Hospital
Acronym: LANA
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0483; 2024-A1986-41 (Other: ANSM)
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leucemia; High-risk Myelodysplastic Syndrome (MDS); Acute Lymphoid Leukemia
Keywords: high-risk myelodysplactic syndrome; Acute leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bone narrow samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with high-risk AML, ALL or MDS: Patients with high-risk AML, ALL or MDS treated in the hematology department of Nantes University Hospital.
  According to the needs of ongoing biological studies, additional volumes may be collected during blood and bone marrow sampling for diagnosis or relapse at inclusion , with up to one additional sample each month for three months following inclusion

SUMMARY:
The aim of the LANA bio-collection is to collect samples from patients with Acute Myeloid Leukemia (AML), Acute Lymphocytic Leukemia (ALL) or or high-risk myelodysplastic syndrome (MDS) to facilitate access to the leukemic or myelodysplastic cells for the research teams of the National Institute of Health and Medical Research (INSERM). To do this, an additional blood or bone marrow sample to those planned in the context of patient care will be collected after signing consent. These samples will then be sent directly to the INSERM teams for immediate analysis with the aim to conduct research aimed at a better understanding of AML, ALL or MDS and improving treatments

DETAILED DESCRIPTION:
The main objective of the prospective and monocentric LANA biocollection is to characterize the tumor and its microenvironment in Acute Lymphocytic Leukemia (ALL) or Acute Myeloid Leukemia (AML) or high-risk myelodysplastic syndrome (MDS) in order to identify new biomarkers or therapeutic targets. Blood and bone marrow of patients included in the LANA bio-collection will be used to search for genetic polymorphisms linked to an increased risk of developing AML or ALL and on the analysis of the evolution of plasma concentrations of a wide range of cytokines. This approach will involve an in-depth study of their transcriptome, followed by the validation of cell populations and potential therapeutic targets by multiparametric flow cytometry on fresh samples.

The LANA bio-collection will be proposed by a physician to patients regardless of the stage of the disease. The inclusion in the biocollection will be effective following the signing of the consent form. An additional volume of blood and bone marrow samples will be taken only if these sampling are already planned in the patient care and without any additional puncture being performed. Sampling will not be taken on a recurring basis but, according to the needs of ongoing biological studies, additional samples may be collected, with up to one additional sample each month for three months following inclusion. Blood and bone marrow samples will be taken at the time of inclusion (for diagnosis or relapse) and, based on the results of the first analyses of the laboratories of research partners, it is possible that the biological materials available in the initial samples are not sufficient to continue the explorations. In this case, the laboratory will contact the clinic service for a new addition of blood or medullary samples collected during patient care. The collected samples will either be sent directly to the partner research laboratories or, if not sent immediately, will be stored in the laboratory dedicated to clinical research sample processing within the clinical hematology department of Nantes University Hospital, under the responsibility of the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age affected by AML, ALL or MDS regardless of the time of treatment
* Patient who has signed the consent form.
* Patient affiliated with a social security system.

Exclusion Criteria:

* Minor patients.
* Adults under guardianship.
* Protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk AML, ALL, or MDS managed in the hematology department of the University Hospital of Nantes
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2034-11-15 (Estimated); Study Completion 2034-11-15 (Estimated)

PRIMARY OUTCOMES:
Characterization of the tumor and its microenvironment for AML, ALL or MDS in order to identify novel biomarkers or therapeutic targets | One year after inclusion
  Identify genetic polymorphisms associated with an increased risk of developing AML or ALL

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Peterlin, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided